CLINICAL TRIAL: NCT00974298
Title: Uncemented Total Elbow Arthroplasty Data Collection
Status: Terminated | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Donald Lee, Professor of Orthopaedic Surgery, Vanderbilt University
Other Study IDs: 090342
Record Dates: First submitted 2009-09-02; First posted 2009-09-10 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Total Elbow Arthroplasty
MeSH Terms: interventions — Arthroplasty, Replacement, Elbow

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Elbow replacement: There are no other arms other then an uncemented total elbow replacement.
  Interventions: Procedure: Total elbow replacement arthroplasty

INTERVENTIONS:
Procedure: Total elbow replacement arthroplasty — Total elbow arthroplasty using pressfit technique in which no cement is used.

SUMMARY:
The purpose of this study is to document the performance and clinical outcomes of uncemented total elbow replacements involving the press-fit technique performed at the Vanderbilt Hand Center. The press-fit use technique is often used because of complications with cement loosening.

DETAILED DESCRIPTION:
The three parts of this study will be:

Retrospective Chart Review-

A chart review will be completed on all patients that have had an uncemented total elbow arthroplasty using the press-fit technique at Vanderbilt Hand & Upper Extremity Center. The chart review will include:

* A historical data form
* An operative data form
* A radiographic assessment form

Questionnaire Mailing- We will mail prospective study patients a DASH (Disabilities of the Arm, Shoulder and Hand) questionnaire to complete with a mailing letter explaining the request for this information. The DASH will be modified to ask patients regarding their pre-operative time as well.

Clinical Data Collection-

We will enroll patients who have already had/or will be having a uncemented total elbow arthroplasty using the press-fit technique. If the patient already has a file completed through the chart review we will not complete the historical data form, operative form, or previous radiograph assessments. If the patient does not have a file completed through the chart review the data collection will include:

* An Informed Consent Document
* A historical data form
* An operative data form
* A radiographic assessment form
* Patient-completed DASH questionnaire
* Elbow Assessment Form

ELIGIBILITY:
Inclusion Criteria:

* Any patient who has had a total elbow arthroplasty using a press-fit technique at the Vanderbilt Hand & Upper Extremity Center

Exclusion Criteria:

* Patients less than 18 years old
* For chart review and post-operative enrollment the patients must have adequate radiographs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who require total elbow arthroplasty.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2009-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Patient examination measurements and radiographic measurements will be used to determine the effects of an uncemented total elbow arthroplasty | Pre-operative to five year post-operative appointment

CONTACTS AND LOCATIONS:
Overall Officials: Donald Lee, M.D., Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Hand & Upper Extremity Center, Nashville, Tennessee, United States